CLINICAL TRIAL: NCT01592773
Title: An Open-Label Extension Study of the Safety and Tolerability of Memantine in Pediatric Patients With Autism, Asperger's Disorder, or Pervasive Developmental Disorder Not Otherwise Specified (PDD-NOS)
Brief Title: Safety Study of Memantine in Pediatric Patients With Autism, Asperger's Disorder or Pervasive Developmental Disorder Not Otherwise Specified (PDD-NOS)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated because primary efficacy parameter failed to demonstrate statistically significant difference between memantine and placebo in controlled trials
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEM-MD-69
Record Dates: First submitted 2012-05-03; First posted 2012-05-07 (Estimated); Results first posted 2015-02-16 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-01

CONDITIONS: Autism Spectrum Disorder (ASD); Autism; Autistic Disorder; Asperger's Disorder; Asperger's; Pediatric Autism; Pervasive Developmental Disorder Not Otherwise Specified (PDD-NOS)
Keywords: Autistic Disorder; Asperger's Disorder; Asperger's; Pediatric Autism; Pervasive Developmental Disorder Not Otherwise Specified (PDD-NOS); Pervasive Child Development Disorder
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Asperger Syndrome | interventions — Memantine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Memantine (Experimental): To maintain the blind of the preceding study, patients who participated in MEM-MD-68 (NCT01592747) began this study with 6 weeks of double blind dosing during which all patients were either titrated to or remained on their maximum target dosages. This was followed by up-to 42 weeks of open-label dosing.
  Patients who took open-label memantine in study MEM-MD-67 (NCT01999894) or MEM-MD-91(NCT01592786), received up to 48 weeks of open-label memantine at their maximum tolerated weight based target dosage.
  Interventions: Drug: Memantine Hydrochloride (HCl)

INTERVENTIONS:
Drug: Memantine Hydrochloride (HCl) — During the 6-week double-blind dosing titration/maintenance period, Memantine extended-release 3-mg and 6-mg capsules; oral administration. Dosing was once daily.
  During open-label treatment: Memantine extended-release 3mg capsules; oral administration. The maximum target dosage was identified during the prior studies for each patient. Dosing was once daily.
  Other Names: Namenda

SUMMARY:
The objective of this study is to evaluate the long-term safety and tolerability of memantine in the treatment of pediatric patients with autism, Asperger's Disorder or Pervasive Developmental Disorder Not Otherwise Specified (PDD-NOS).

DETAILED DESCRIPTION:
This clinical study was a 48-week, multicenter, multinational, open-label extension study in pediatric outpatients with autism, Asperger's Disorder, or PDD-NOS conducted at 106 study centers. Patients were eligible for this long-term extension study if they had:

* completed the open-label Study MEM MD 67,or
* completed the open-label Study MEM-MD-91, or
* completed the double-blind Study MEM-MD-68, or
* discontinued study MEM-MD-68 by meeting requirements for loss of therapeutic response

The weight-based dose limits in this study were as follows:

Group A: ≥ 60 kg; maximum 15 mg/day Group B: 40-59 kg; maximum 9 mg/day Group C: 20-39 kg; maximum 6 mg/day Group D: < 20 kg; maximum 3 mg/day

The decision to close the study early was based on data from 2 double-blind placebo-controlled studies (MEM-MD-57A and MEM-MD-68) that failed to demonstrate a statistically significant difference between memantine and placebo in the primary efficacy parameter based on Social Responsiveness Scale (SRS) total raw score.

ELIGIBILITY:
Inclusion Criteria:

* Patients who completed Study MEM-MD-67, MEM-MD-68, MEM-MD-91, or discontinued Study MEM-MD-68 due to meeting the criterion for loss of therapeutic response.
* Having normal results from a physical examination and laboratory tests at Visit 1 of this study (last visit of the preceding study). Any abnormal findings must be deemed not clinically significant by the Investigator and documented as such.
* Have a family that is sufficiently organized and stable to guarantee adequate safety monitoring and continuous attendance to clinic visits for the duration of the study

Exclusion Criteria:

* Patients who discontinued a preceding memantine study due to an adverse event possibly related to study drug
* Patients with a concurrent medical condition that might interfere with the conduct of the study, confound interpretation of the study results, or endanger the patient's well being
* Significant risk of suicidality based on the Investigator's judgment, Aberrant Behavior Checklist-irritability subscale (ABC-I), or if appropriate, as indicated by a response of "yes" to questions 4 or 5 in the suicidal ideation section of the Children's Columbia-Suicide Severity Rating Scale (C-SSRS) or any suicidal behavior

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 747 (Actual)
Dates: Start 2012-10; Primary Completion 2014-01 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Lateiner, MS, MBA, Study Director — Forest Research Institute, Inc.- A Subsidiary of Forest Laboratories, Inc.
Locations (106):
- United States (68):
  - Forest Investigative Site 068, Dothan, Alabama
  - Forest Investigative Site 005, Phoenix, Arizona
  - Forest Investigative Site 055, Tucson, Arizona
  - Forest Investigative Site 077, Little Rock, Arkansas
  - Forest Investigative Site 054, Glendale, California
  - Forest Investigative Site 109, Imperial, California
  - Forest Investigative Site 066, Irvine, California
  - Forest Investigative Site 096, Los Angeles, California
  - Forest Investigative Site 021, San Francisco, California
  - Forest Investigative Site 026, Santa Ana, California
  - Forest Investigative Site 002, Stanford, California
  - Forest Investigative Site 078, Boulder, Colorado
  - Forest Investigative Site 073, Centennial, Colorado
  - Forest Investigative Site 052, Washington D.C., District of Columbia
  - Forest Investigative Site 075, Bradenton, Florida
  - Forest Investigative Site 080, Gainesville, Florida
  - Forest Investigative Site 117, Jacksonville, Florida
  - Forest Investigative Site 065, Maitland, Florida
  - Forest Investigative Site 118, Miami, Florida
  - Forest Investigative Site 085, Oakland Park, Florida
  - Forest Investigative Site 115, Orange City, Florida
  - Forest Investigative Site 125, Orlando, Florida
  - Forest Investigative Site 062, Orlando, Florida
  - Forest Investigative Site 067, Tampa, Florida
  - Forest Investigative Site 101, Wellington, Florida
  - Forest Investigative Site 102, Libertyville, Illinois
  - Forest Investigative Site 023, Naperville, Illinois
  - Forest Investigative Site 082, Evansville, Indiana
  - Forest Investigative Site 123, Fort Wayne, Indiana
  - Forest Investigative Site 056, Indianapolis, Indiana
  - Forest Investigative Site 061, Louisville, Kentucky
  - Forest Investigative Site 095, Lake Charles, Louisiana
  - Forest Investigative Site 091, New Orleans, Louisiana
  - Forest Investigative Site 086, Rockville, Maryland
  - Forest Investigative Site 059, Newton, Massachusetts
  - Forest Investigative Site 108, Springfield, Massachusetts
  - Forest Investigative Site 116, Lincoln, Nebraska
  - Forest Investigative Site 097, Lincoln, Nebraska
  - Forest Investigative Site 130, Henderson, Nevada
  - Forest Investigative Site 104, Las Vegas, Nevada
  - Forest Investigative Site 136, Neptune City, New Jersey
  - Forest Investigative Site 127, Toms River, New Jersey
  - Forest Investigative Site 081, Albuquerque, New Mexico
  - Forest Investigative Site 107, Albuquerque, New Mexico
  - Forest Investigative Site 098, The Bronx, New York
  - Forest Investigative Site 072, Chapel Hill, North Carolina
  - Forest Investigative Site 069, Avon Lake, Ohio
  - Forest Investigative Site 001, Columbus, Ohio
  - Forest Investigative Site 019, Oklahoma City, Oklahoma
  - Forest Investigative Site 092, Tulsa, Oklahoma
  - Forest Investigative Site 053, Gresham, Oregon
  - Forest Investigative Site 132, Johnstown, Pennsylvania
  - Forest Investigative Site 131, McMurray, Pennsylvania
  - Forest Investigative Site 100, Media, Pennsylvania
  - Forest Investigative Site 105, Charleston, South Carolina
  - Forest Investigative Site 090, Memphis, Tennessee
  - Forest Investigative Site 057, Nashville, Tennessee
  - Forest Investigative Site 051, Houston, Texas
  - Forest Investigative Site 070, The Woodlands, Texas
  - Forest Investigative Site 028, Clinton, Utah
  - Forest Investigative Site 141, Ogden, Utah
  - Forest Investigative Site 029, Salt Lake City, Utah
  - Forest Investigative Site 064, Charlottesville, Virginia
  - Forest Investigative Site 113, Norfolk, Virginia
  - Forest Investigative Site 124, Roanoke, Virginia
  - Forest Investigative Site 071, Bothell, Washington
  - Forest Investigative Site 119, Charleston, West Virginia
  - Forest Investigative Site 063, Middleton, Wisconsin
- Belgium (2):
  - Forest Investigative Site 204, Brussels
  - Forest Investigative Site 203, Jette
- Forest Investigative Site 155, Toronto, Ontario, Canada
- Colombia (3):
  - Forest Investigative Site 228, Antioquia, Bello
  - Forest Investigative Site 227, Barranquilla
  - Forest Investigative Site 226, Bogotá
- Forest Investigative Site 276, Tallinn, Estonia
- Forest Investigative Site 329, Bron, Rhone, France
- Hungary (4):
  - Forest Investigative Site 381, Budapest
  - Forest Investigative Site 376, Budapest
  - Forest Investigative Site 378, Budapest
  - Forest Investigative Site 382, Gyula
- Forest Investigative Site 401, Kopavogur, Iceland
- Italy (2):
  - Forest Investigative Site 453, Roma
  - Forest Investigative Site 452, Siena
- Forest Investigative Site 526, Wellington, New Zealand
- Poland (5):
  - Forest Investigative Site 579, Gdansk
  - Forest Investigative Site 578, Gdansk
  - Forest Investigative Site 580, Kielce
  - Forest Investigative Site 576, Tyniec Mały
  - Forest Investigative Site 577, Warsaw
- Serbia (4):
  - Forest Investigative Site 626, Belgrade
  - Forest Investigative Site 627, Belgrade
  - Forest Investigative Site 629, Niš
  - Forest Investigative Site 628, Novi Sad
- Forest Investigative Site 676, Bellville Cape Town, South Africa
- South Korea (4):
  - Forest Investigative Site 704, Yangsan, Gyeongsangnam-do
  - Forest Investigative Site 702, Seoul
  - Forest Investigative Site 703, Seoul
  - Forest Investigative Site 701, Seoul
- Spain (3):
  - Forest Investigative Site 729, Barcelona
  - Forest Investigative Site 728, Sabadell
  - Forest Investigative Site 730, Torremolinos
- Ukraine (5):
  - Forest Investigative Site 803, Donetsk
  - Forest Investigative Site 807, Kharkiv
  - Forest Investigative Site 802, Kherson
  - Forest Investigative Site 804, Kyiv
  - Forest Investigative Site 801, Odesa

REFERENCES:
- [Derived] Brignell A, Marraffa C, Williams K, May T. Memantine for autism spectrum disorder. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013845. doi: 10.1002/14651858.CD013845.pub2. PMID 36006807

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient recruitment occurred over an eleven month period, from October of 2012 to September of 2013, at 106 study sites, located in the United States and 15 other countries.
Groups:
- Memantine: To maintain the blind of the preceding study, patients who participated in MEM-MD-68 began this study with 6 weeks of double blind dosing during which all patients were either titrated to or remained on their maximum target dosages. This was followed by up-to 42 weeks of open-label dosing.
  Patients who took open-label memantine in the preceding study, MEM-MD-67 or MEM-MD-91, received up to 48 weeks of open-label memantine at their maximum tolerated weight based target dosage.
Period: Overall Study
Arm/Group | Memantine
Started | 747 (All enrolled patients received at least 1 dose of investigational product (Safety Population).)
Completed | 81
Not Completed | 666
Not completed — Study Terminated by Sponsor | 582
Not completed — Withdrawal by Subject | 35
Not completed — Lost to Follow-up | 19
Not completed — Adverse Event | 17
Not completed — Lack of Efficacy | 9
Not completed — Protocol Violation | 2
Not completed — Inclusion/exclusion not meet | 1
Not completed — Other Reason | 1

BASELINE CHARACTERISTICS:
Population: Demographic summaries were provided based on the 747 patients who received at least 1 dose of investigational product in the extension study (Safety Population).
Arm/Group | Memantine
Number analyzed (Participants) | 747
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.0 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120
  Male | 627
Race/Ethnicity, Customized [Number; unit: participants]
  White | 636
  Black or African American | 42
  Asian | 44
  American Indian or Alaska Native | 2
  Native Hawaiian or Other Pacific Islander | 3
  Other Race | 20
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 88
  Not Hispanic or Latino | 659
Region of Enrollment [Number; unit: participants]
  United States | 586
  Belgium | 4
  Canada | 1
  Colombia | 8
  Estonia | 5
  France | 9
  Hungary | 14
  Iceland | 5
  Italy | 6
  Korea, Republic of | 22
  New Zealand | 1
  Poland | 36
  Serbia | 21
  South Africa | 1
  Spain | 14
  Ukraine | 14

OUTCOME MEASURES:

1. Primary Outcome: Patients With Any Treatment-emergent Adverse Event
Description: Number of patients who experienced 1 or more Treatment Emergent Adverse Event
Time Frame: Visit 1 (Week 0) up to 30 days after Visit 8 (up to Week 48) or Final Visit
Population: Analysis was performed on the 747 patients who took at least 1 dose of investigational product (Safety Population).
Measure: Number; unit: participants
Arm/Group | Memantine
Number analyzed (Participants) | 747
participants | 424

ADVERSE EVENTS:
Time Frame: Adverse Event data was collected from October 2012 to February 2014 at 106 sites in the US and 15 other countries.
Description: Safety results are based on the safety population (ie, all patients who took at least one dose of investigational product).
Arm/Group | Memantine
Serious Adverse Events (participants affected / at risk) | 8/747
Other Adverse Events (participants affected / at risk) | 150/747
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Memantine (N=747)
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain lower (Gastrointestinal disorders) | 1
Abnormal behaviour (Nervous system disorders) | 1
Appendicitis (Infections and infestations) | 1
Dehydration (Investigations) | 1
Dysphoria (Nervous system disorders) | 1
Foreign body (Injury, poisoning and procedural complications) | 1
Homicidal ideation (Nervous system disorders) | 1
Rectal prolapse (Injury, poisoning and procedural complications) | 1
Suicidal ideation (Nervous system disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Memantine (N=747)
Vomiting (Gastrointestinal disorders) | 51
Pyrexia (General disorders) | 47
Nasopharyngitis (Infections and infestations) | 55
Headache (Nervous system disorders) | 41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated in this study will be the property of Forest Research Institute, Inc. An integrated clinical and statistical report will be prepared at the completion of the study.

Publication of the results by the PI will be subject to mutual agreement between the PI and Forest Research Institute, Inc.